CLINICAL TRIAL: NCT01092845
Title: Double-Blind, Randomized, Multiple-Dose, Placebo-Controlled, 2-Way Crossover Study To Study Effects of PF-04457845 On Polysomnographic Endpoints In Healthy Volunteers
Brief Title: Study To Establish The Effects Of PF-04457845 On Sleep In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: B0541010
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Healthy; Sleep
Keywords: Double-Blind; Randomized; Placebo-Controlled; 2-Way Crossover; Polysomnographic Endpoints
MeSH Terms: interventions — N-pyridazin-3-yl-4-(3-((5-(trifluoromethyl)pyridin-2-yl)oxy)benzylidene)piperidine-1-carboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-04457845 followed by placebo (Experimental)
  Interventions: Drug: PF-04457845 / matched placebo
- Placebo followed by PF-04457845 (Experimental)
  Interventions: Drug: PF-04457845 / matched placebo

INTERVENTIONS:
Drug: PF-04457845 / matched placebo — PF-04457845 4 mg tablet once daily / matched placebo
  Arms: PF-04457845 followed by placebo
Drug: PF-04457845 / matched placebo — PF-04457845 4 mg tablet once daily / matched placebo
  Arms: Placebo followed by PF-04457845

SUMMARY:
PF-04457845 has been shown to temporarily decrease the dream (REM) period of sleep in rats, which suggests that PF-04457845 is active in rat's brains. This study is designed to see whether this is also the case in man.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 and 55 years
* Body Mass Index (BMI) between 17.5 and 30.5 kg/m2
* Total body weight >50 kg

Exclusion Criteria:

* History of any active sleep disorder
* History of any sleep or circadian rhythm sleep disorder including RLS, narcolepsy, sleep apnea, phase advance or delay syndromes within the past 5 years
* Currently on or planning to be involved in night or rotating shift work or traveling across more than four time zones in 14 days prior to screening

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Percentage of total sleep time spent in REM (ie, time spent in REM/total sleep time) | 3 days

SECONDARY OUTCOMES:
Minutes of REM sleep time | 3 days
Percentage of total sleep time spent in Stage 1 sleep | 3 days
Percentage of total sleep time spent in Stage 2 sleep | 3 days
Percentage of total sleep time spent in Stage 3-4 sleep | 3 days
Total sleep time | 3 days
Wake after sleep onset (sum of wake time during sleep and prior to final awakening) and wake time after sleep) (WASO) | 3 days
Number of arousals after sleep onset (NASO) | 3 days
Latency to persistent sleep | 3 days
Plasma concentrations of PF-04457845 | 3 days
Plasma concentrations of fatty acid amides (N-arachidonyl ethanolamine (anandamide, AEA), palmitoylethanolamide (PEA), oleoylethanolamide (OEA) and linoleoyl ethanolamine (LEA)) | 3 days
Beta-band spectral power (qEEG) measured with eyes open and eyes closed while subjects are awake immediately before lights off for each PSG | 3 days
Beta-band spectral power (qEEG) measured with eyes open and eyes closed while subjects are awake immediately after lights on for each PSG | 3 days
Beta-band spectral power (qEEG) measured while subjects are asleep during the sleep onset period (SOP) and first 3 periods of NREM sleep | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New York, New York, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0541010&StudyName=Study%20To%20Establish%20The%20Effects%20Of%20PF-04457845%20On%20Sleep%20In%20Healthy%20Volunteers